CLINICAL TRIAL: NCT04015388
Title: Development of a Comprehensive Clinical Decision Support System and Educational Tool to Support Optimization of Glycemic Control in the Hospital and Critical Care Setting
Brief Title: Optimization of Glycemic Control in the Hospital and Critical Care Setting
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Ravi Tripathi, Principal Investigator, Clinical Assistant Professor, Ohio State University
Other Study IDs: 2013H0285
Record Dates: First submitted 2019-07-06; First posted 2019-07-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Hyperglycemia; Diabetes Mellitus
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Diabetes Mellitus / Hyperglycemia: iPro Continuous Glucose Monitoring on subjects with blood sugar value >140 mg/dL upon admission to the intensive care unit or who have been diagnosed with type 1 or type 2 diabetes or have glycosylated hemoglobin A1C (HbA1C) values > 6.5% prior to admission.
  Interventions: Device: iPro Continuous Glucose Monitoring

INTERVENTIONS:
Device: iPro Continuous Glucose Monitoring — iPro device is a continuous glucose monitoring (CGM) FDA approved device. This CGM device consists of a small recorder which reports glucose values every five minutes. This recorder is connected directly to a glucose sensor. The glucose-oxidase based sensor measures extracellular fluid in the subcutaneous tissue. The tiny and flexible sensors are typically inserted just beneath the skin, usually in the abdominal area, but can also be placed in the buttock, or anterior or lateral thigh.

SUMMARY:
Continuous Glucose Monitoring collected using the iPro device, to complete a large dataset consisting of routine electronic health records, biological, neurophysiological, physiological, and glycemic data. This dataset will eventually contribute to the further development and optimization of a comprehensive simulation, training, and clinical decision support system designed to contribute the optimization of glycemic control in the hospital and critical care setting.

DETAILED DESCRIPTION:
Although recent advances in technology such as electronic medical records and continuous glucose monitoring provide enhanced monitoring capabilities, optimal glycemic control in the hospital and critical care setting is still extremely difficult to obtain. These technologies provide little to no identification of trends in data, and clinical decision support.

The goal of this research study was to collect data to support further development and optimization of a comprehensive clinical decision support system with simulation, training, and clinical decision support functionality. The system will also be designed to provide real-time performance measurement and feedback to ensure glycemic control is maintained at an optimal level.

The continuous glucose monitor (CGM) device utilized in this investigation was the iPro Recorder® (Medtronic Diabetes, Northridge, CA), a FDA approved monitoring device which reports glucose values every five minutes.

Subjects with a history of hyperglycemia or current hyperglycemia were identified either in the intensive care unit or prior to surgery. Upon enrollment of eligible patients in the study, CGM device was placed on subject's abdomen or thigh. The times logged by the CGM device were synchronized to achieve valid data pairing according to time. Subjects were visited as needed or at least twice in a 24-hour period to ensure that the devices were still in place and comfortable for the patient. After 72 hours of data collection, the CGM device was removed and the area of attachment cleaned.

Research staff collected medical history and standard of care glucose point of care obtained during subject's participation into the study. Other data from the patient's standard of care monitor, such as oxygen saturation levels, blood pressure, respiratory and heart rate, were collected as part of the patient's safety assessment assurance.

Data analysis will be completed offsite by investigators at Aptima, Inc. and their wholly owned subsidiary, Analytic Diabetic Systems, LLC. All patient data collected in this investigation was appropriately de-identified.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, ≥ 18 years of age.
2. Subject able to provide written informed consent to participate in the study.
3. Female subject with a negative urine or serum pregnancy test, or not of childbearing potential, defined as surgically sterile due to bilateral tubal ligation, bilateral oophorectomy or hysterectomy; or are postmenopausal for at least 1 year.
4. Have a blood sugar value of >140 mg/dL or an glycosylated hemoglobin A1C (HbA1C) values >6.5% upon admission to the surgical Intensive Care Unit (ICU), medical ICU, or cardiovascular ICU, and have or not have been diagnosed with type 1 or type 2 diabetes.

Exclusion Criteria:

1. Subjects younger than 18 years old.
2. Subjects who are prisoners.
3. Subjects with known hypersensitivity to latex or tape.
4. Females who are pregnant or breastfeeding.
5. Subjects unable to provided informed consent.
6. Subjects unable to participate in the study for any reason in the opinion of the Principal Investigator.
7. Subjects enrolled in other research studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population included in this study were adult patients, with at least 18 years old, admitted in The Ohio State University Wexner Medical Center critical care setting. Subjects had a blood sugar value >140 mg/dL upon admission to ICU or had been diagnosed with type 1 or type 2 diabetes or had glycosylated hemoglobin A1C (HbA1C) values > 6.5% prior to admission.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2014-08-19 (Actual); Primary Completion 2016-08-02 (Actual); Study Completion 2021-02-04 (Actual)

PRIMARY OUTCOMES:
Evaluate performance of glucose predictive models, clinical decision support algorithms, and performance measures in simulated real-time setting. | Glucose levels collected since placement of the iPro device (Hour 0) until removal of the ipro device (Hour 72)
  Glucose measurements collected (mg/dL) in the iPro device will be further analyzed to create an algorithm to predict glucose changes (hyperglycemia or hypoglycemia).

SECONDARY OUTCOMES:
Ensure data collected has considerable quantity of hypoglycemia, normoglycemia, and hyperglycemia for algorithm model development and optimization. | Glucose levels collected since placement of the iPro device (Hour 0) until removal of the ipro device (Hour 72)
  Glucose measurements collected (mg/dL) in the iPro device will be reviewed to confirmed that sufficient hyperglycemia or hypoglycemia episodes, as well as normal glucose values, were recorded. Available data will be used to create the algorithm to predict glucose changes.
Further development of GlyCU system functionality (simulation, training, and clinical decision support capabilities) and identification of necessary steps for integration with the OSUWMC electronic health record database. | Glucose levels collected since placement of the iPro device (Hour 0) until removal of the ipro device (Hour 72)
  Correlate glucose measurements collected (mg/dL) in the iPro device with the glucose values collected as at standard of care for each study subject at the Ohio State University Wexner Medical Center (OSUWMC).

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Tripathi, MD, Principal Investigator — Ohio State University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cox DJ, Gonder-Frederick LA, Kovatchev BP, Julian DM, Clarke WL. Progressive hypoglycemia's impact on driving simulation performance. Occurrence, awareness and correction. Diabetes Care. 2000 Feb;23(2):163-70. doi: 10.2337/diacare.23.2.163. PMID 10868825
- [Background] Engoren M, Schwann TA, Habib RH. Elevated hemoglobin A1c is associated with readmission but not complications. Asian Cardiovasc Thorac Ann. 2014 Sep;22(7):800-6. doi: 10.1177/0218492313515895. Epub 2013 Dec 6. PMID 24887924
- [Background] Giugliano D, Marfella R, Coppola L, Verrazzo G, Acampora R, Giunta R, Nappo F, Lucarelli C, D'Onofrio F. Vascular effects of acute hyperglycemia in humans are reversed by L-arginine. Evidence for reduced availability of nitric oxide during hyperglycemia. Circulation. 1997 Apr 1;95(7):1783-90. doi: 10.1161/01.cir.95.7.1783. PMID 9107164
- [Background] Ingels C, Debaveye Y, Milants I, Buelens E, Peeraer A, Devriendt Y, Vanhoutte T, Van Damme A, Schetz M, Wouters PJ, Van den Berghe G. Strict blood glucose control with insulin during intensive care after cardiac surgery: impact on 4-years survival, dependency on medical care, and quality-of-life. Eur Heart J. 2006 Nov;27(22):2716-24. doi: 10.1093/eurheartj/ehi855. Epub 2006 Apr 11. PMID 16608860
- [Background] Inzucchi SE, Siegel MD. Glucose control in the ICU--how tight is too tight? N Engl J Med. 2009 Mar 26;360(13):1346-9. doi: 10.1056/NEJMe0901507. Epub 2009 Mar 24. No abstract available. PMID 19318385
- [Background] Kanji S, Buffie J, Hutton B, Bunting PS, Singh A, McDonald K, Fergusson D, McIntyre LA, Hebert PC. Reliability of point-of-care testing for glucose measurement in critically ill adults. Crit Care Med. 2005 Dec;33(12):2778-85. doi: 10.1097/01.ccm.0000189939.10881.60. PMID 16352960
- [Background] Sung J, Bochicchio GV, Joshi M, Bochicchio K, Tracy K, Scalea TM. Admission hyperglycemia is predictive of outcome in critically ill trauma patients. J Trauma. 2005 Jul;59(1):80-3. doi: 10.1097/01.ta.0000171452.96585.84. PMID 16096543
- [Background] Van den Berghe G. How does blood glucose control with insulin save lives in intensive care? J Clin Invest. 2004 Nov;114(9):1187-95. doi: 10.1172/JCI23506. PMID 15520847
- [Background] Pappada SM, Borst MJ, Cameron BD, Bourey RE, Lather JD, Shipp D, Chiricolo A, Papadimos TJ. Development of a neural network model for predicting glucose levels in a surgical critical care setting. Patient Saf Surg. 2010 Sep 9;4(1):15. doi: 10.1186/1754-9493-4-15. PMID 20828400
- [Background] Pappada SM, Cameron BD, Tulman DB, Bourey RE, Borst MJ, Olorunto W, Bergese SD, Evans DC, Stawicki SP, Papadimos TJ. Evaluation of a model for glycemic prediction in critically ill surgical patients. PLoS One. 2013 Jul 19;8(7):e69475. doi: 10.1371/journal.pone.0069475. Print 2013. PMID 23894489